CLINICAL TRIAL: NCT01657279
Title: Clinician JUdgment Versus Risk Score to Predict Stroke outComes:
Brief Title: Clinician JUdgment Versus Risk Score to Predict Stroke outComes: The JURASSIC Clinical Trial
Acronym: JURASSIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Gustavo Saposnik, Staff Physician and Clinician Scientist, Associate Professor of medicine, University of Toronto, Unity Health Toronto
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: SMH 09-020; 09-020 (Other: St Michael's Hospital, University of Toronto)
Record Dates: First submitted 2012-07-30; First posted 2012-08-06 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Stroke; Ischemic Stroke; Cerebrovascular Disease
Keywords: stroke; risk score; iScore; outcomes; mortality; disability; institutionalization
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Randomized clinical scenarios (Experimental): Clinicians are randomized to a sequence of 5 clinical scenarios
  Interventions: Other: Clinical scenarios

INTERVENTIONS:
Other: Clinical scenarios — Clinicians will be randomized to a sequence of 5 clinical scenarios with a variable range of expected outcome [i.e. from low (<10%) to high (>50%) expected risk death at 30 days].

SUMMARY:
Background: Several risk score models are now available to assist clinicians estimate outcomes after an acute ischemic stroke. Limited information is available on the predictive value of these scores compared to real outcomes and clinical judgment.

Objectives: To compare clinician judgment with the use of a validated stroke risk score (iScore) and patients' outcomes.

DETAILED DESCRIPTION:
A convenience sample of 111 practicing clinicians (general and vascular neurologists, internists, and ER physicians) predicted the outcomes of 5 stroke patients based on case summaries. Cases were randomly selected as being representative of the 10 most common clinical scenarios (n=1,415) from a pool of over 12,000 patients admitted to stroke centers in Ontario, Canada. Stroke cases had known clinical presentation, comorbidities, stroke severity, and outcomes.

All participants are active practicing physicians caring for patients with acute stroke. Conditions were standardized to mimic clinical practice.

Main outcomes of interest included 30-day mortality and death or disability at discharge.

Secondary outcome: death or institutionalization at discharge

ELIGIBILITY:
Inclusion Criteria:

* Practicing and active physicians managing patients with stroke

Exclusion Criteria:

* retired physicians
* physicians not exposed to care for stroke patients

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
30 Day Mortality or Disability (mRS >3) at discharge | Death after 30 days from ischemic stroke onset or Disability following hospital discharge

SECONDARY OUTCOMES:
Death at 30 days | 30 days
Death or institutionalization at discharge | up to 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Saposnik, MD MSc FRCPC, Principal Investigator — Unity Health Toronto
Locations (4):
- Duke University Medical Center, Durham, North Carolina, United States
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Background] Saposnik G, Fang J, Kapral MK, Tu JV, Mamdani M, Austin P, Johnston SC; Investigators of the Registry of the Canadian Stroke Network (RCSN); Stroke Outcomes Research Canada (SORCan) Working Group. The iScore predicts effectiveness of thrombolytic therapy for acute ischemic stroke. Stroke. 2012 May;43(5):1315-22. doi: 10.1161/STROKEAHA.111.646265. Epub 2012 Feb 3. PMID 22308252
- [Background] Saposnik G, Raptis S, Kapral MK, Liu Y, Tu JV, Mamdani M, Austin PC; Investigators of the Registry of the Canadian Stroke Network and the Stroke Outcome Research Canada Working Group. The iScore predicts poor functional outcomes early after hospitalization for an acute ischemic stroke. Stroke. 2011 Dec;42(12):3421-8. doi: 10.1161/STROKEAHA.111.623116. Epub 2011 Sep 29. PMID 21960583
- [Background] Saposnik G, Kapral MK, Liu Y, Hall R, O'Donnell M, Raptis S, Tu JV, Mamdani M, Austin PC; Investigators of the Registry of the Canadian Stroke Network; Stroke Outcomes Research Canada (SORCan) Working Group. IScore: a risk score to predict death early after hospitalization for an acute ischemic stroke. Circulation. 2011 Feb 22;123(7):739-49. doi: 10.1161/CIRCULATIONAHA.110.983353. Epub 2011 Feb 7. PMID 21300951
- See also: Web based tool for estimating outcomes using the iScore to compare clinicians' estimations — http://www.sorcan.ca/iscore/